CLINICAL TRIAL: NCT00980174
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Study to Compare the Efficacy and Safety of Denosumab Versus Placebo in Males With Low Bone Mineral Density
Brief Title: Study to Compare the Efficacy and Safety of DenosumAb Versus Placebo in Males With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20080098
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Low Bone Mass; Low Bone Mineral Density; Males With Osteoporosis; Osteopenia; Osteoporosis
Keywords: men; male; denosumab; BMD; lumbar spine; ADAMO; The ADAMO Trial; male osteoporosis; osteoporosis in men; males with low bone mineral density
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Multiple Endocrine Neoplasia Type 1 | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Subjects will receive placebo for denosumab (SC injection every 6 months) for 1 year (double-blind phase) followed by 60 mg denosumab (SC injection every 6 months) for 1 year (open-label phase)
  Interventions: Drug: 60 mg denosumab; Other: Placebo
- 1 (Experimental): 60 mg denosumab (SC injection every 6 months) for 1 year (double-blind phase) followed by 60 mg denosumab(SC injection every 6 months) for 1 year (open-label phase). These subjects will be on denosumab for a total of 2 years.
  Interventions: Drug: 60 mg denosumab

INTERVENTIONS:
Drug: 60 mg denosumab — 60 mg denosumab (SC injection every 6 months)
  Other Names: denosumab
Other: Placebo — Placebo for denosumab (SC injection every 6 months)
  Arms: 2

SUMMARY:
The purpose of this study is to assess how effective and safe denosumab is in a population of males with low bone mass at risk of fracture. The primary clinical hypothesis is that in men with low bone mineral density, the mean percent change in lumbar spine bone mineral density at 12 months in subjects receiving denosumab will be greater than in subjects receiving placebo. Denosumab is a fully human monoclonal antibody with a high affinity for Receptor Activator of Nuclear Factor (RANK) Ligand that can bind and neutralize the activity of human RANK Ligand similar to the action of endogenous osteoprotegerin.

ELIGIBILITY:
Inclusion Criteria:

* Bone Mineral Density (BMD) values (g/cm2) assessed by the local site at either the lumbar spine OR femoral neck that occur within the ranges specified in the protocol OR For subjects with a history of a major osteoporotic fracture (clinical vertebral, hip, humerus and distal radius fractures) occurring more than 6 months prior to screening, BMD values (g/cm2) assessed by the local site, at either the lumbar spine OR femoral neck that occur within the ranges specified in the protocol.
* At least 2 lumbar vertebrae, at least 1 hip and at least one forearm must be evaluable by Dual X ray Absorptiometry (DXA).
* Ambulatory males 30 to 85 years of age inclusive at the start of screening.
* Provide the appropriate written informed consent before any study specific procedure.

Exclusion Criteria:

* BMD values (g/cm2) as specified in the protocol in subjects with or without a history of major osteoporotic fractures, based on the particular scanner that is used.
* Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
* Any severe or more than 1 moderate vertebral fractures on screening spinal x ray
* Any vertebral fracture diagnosed within the 6 months prior to screening
* Any clinical fracture within the last 6 months prior to screening
* For males with a partner of childbearing potential: Subject refuses to use 2 highly effective methods of contraception for the duration of the study and for 10 months after the last dose of study medication.
* For males with a partner who is pregnant: Subject refuses to use a condom for the duration of the study and for 10 months after the last dose of study medication.
* Previous participation in clinical trials with denosumab or administration of commercial denosumab.
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s).
* Vitamin D deficiency [25(OH) vitamin D level < 20 ng/mL (< 49.9 nmol/L)]. Vitamin D replenishment will be permitted and subjects may be re-screened; see Section 7.
* Hyper- or hypothyroidism; however, stable subjects, in the investigator's opinion, on thyroid hormone replacement therapy are allowed.
* Hyper- or hypoparathyroidism. Intact parathyroid hormone (iPTH) values outside of the reference range as determined by the central laboratory
* Elevated transaminases. Serum aspartate aminotransferase; serum glutamate-oxaloacetic transaminase > 2.5 x upper limit of normal. Serum alanine aminotransferase; serum glutamate pyruvate transaminase > 2.5 x upper limit of normal (both as determined by the central laboratory).
* Significantly impaired renal function as determined by a derived glomerular filtration rate (using the Modification of Diet in Renal Disease formula) of less than or equal to 30 mL/min/1.73 m2 calculated by the central laboratory.
* Hypo- or hypercalcemia based on the central laboratory reference ranges for albumin-adjusted serum calcium.
* Known to have tested positive for human immunodeficiency virus, hepatitis C virus, hepatitis B surface antigen or cirrhosis of the liver.
* Malignancy (except fully resected cutaneous basal cell or squamous cell carcinoma) within the last 5 years.
* Any metabolic bone disease, eg osteomalacia, osteogenesis imperfecta, rheumatoid arthritis, Paget's disease, Cushing's disease or, hyperprolactinemia which may interfere with the interpretation of the findings OR evidence of malabsorption syndromes which might interfere with absorption of vitamin D.
* Received any solid organ or bone marrow transplant or is on chronic immunosuppression for any reason.
* Any laboratory abnormality, which in the opinion of the investigator or Amgen, will prevent the subject from completing the study or interfere with the interpretation of the study results.
* Administration of intravenous bisphosphonate, or fluoride (except for dental treatment) or strontium ranelate.
* Oral bisphosphonate treatment:
* greater than or equal to 3 months cumulatively in the past 2 years, OR
* greater than or equal to 1 month in the past year, OR
* Any use during the 3-month period prior to randomization
* Administration of any of the following treatments 3 months prior to screening:
* Anabolic steroids or testosterone
* Glucocorticosteroids (greater than or equal to 5 mg prednisone equivalent per day for more than 10 days or a total cumulative dose of greater than or equal to 50 mg)
* Calcitonin
* Calcitriol or vitamin D derivatives [vitamin D contained in supplements or multivitamins is allowed]
* Other bone active drugs including anti-convulsives (except benzodiazepines) and heparin
* Chronic systemic ketoconazole, adrenocorticotrophic hormone (ACTH), cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, gonadotropin-releasing hormone agonists.
* Androgen deprivation therapy
* Known sensitivity to mammalian cell derived drug products.
* Known intolerance to calcium or vitamin D supplements.
* Height, weight or girth which may preclude accurate DXA measurements.
* Bilateral hip replacements
* Any physical or psychiatric disorder which, in the opinion of the investigator or Amgen, will prevent the subject from completing the study or interfere with the interpretation of the study results.
* Evidence of alcohol or substance-abuse within the last 12 months which the investigator believes would interfere with understanding of or completion of the study.

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2011-06-21 (Actual); Study Completion 2012-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Langdahl BL, Teglbjaerg CS, Ho PR, Chapurlat R, Czerwinski E, Kendler DL, Reginster JY, Kivitz A, Lewiecki EM, Miller PD, Bolognese MA, McClung MR, Bone HG, Ljunggren O, Abrahamsen B, Gruntmanis U, Yang YC, Wagman RB, Mirza F, Siddhanti S, Orwoll E. A 24-month study evaluating the efficacy and safety of denosumab for the treatment of men with low bone mineral density: results from the ADAMO trial. J Clin Endocrinol Metab. 2015 Apr;100(4):1335-42. doi: 10.1210/jc.2014-4079. Epub 2015 Jan 21. PMID 25607608
- [Background] Orwoll E, Teglbjaerg CS, Langdahl BL, Chapurlat R, Czerwinski E, Kendler DL, Reginster JY, Kivitz A, Lewiecki EM, Miller PD, Bolognese MA, McClung MR, Bone HG, Ljunggren O, Abrahamsen B, Gruntmanis U, Yang YC, Wagman RB, Siddhanti S, Grauer A, Hall JW, Boonen S. A randomized, placebo-controlled study of the effects of denosumab for the treatment of men with low bone mineral density. J Clin Endocrinol Metab. 2012 Sep;97(9):3161-9. doi: 10.1210/jc.2012-1569. Epub 2012 Jun 21. PMID 22723310
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Denosumab 60 mg Q6M
Started | 121 | 121
Completed | 117 | 111
Not Completed | 4 | 10
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Ineligibility determined | 2 | 1
Not completed — Death | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab 60 mg Q6M | Total
Number analyzed (Participants) | 121 | 121 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (9.1) | 64.9 (10.5) | 65.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 121 | 121 | 242
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 107 | 121 | 228
  Hispanic or Latino | 10 | 0 | 10
  Asian | 2 | 0 | 2
  Black or African American | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  Europe | 78 | 87 | 165
  North America | 43 | 34 | 77

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: From Baseline to 12 Months
Population: Subjects with baseline and at least one post baseline measurements
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 118 | 117
Percent | 0.9 [0.3 to 1.4] | 5.7 [5.1 to 6.2]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted by level of baseline bone mineral density T-score; Mean Difference (Net) = 4.8, 95% CI 2-sided [4.0 to 5.6] — Denosumab - Placebo

2. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: From Baseline to 12 Months
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 119 | 117
Percent | 0.3 [-0.1 to 0.7] | 2.4 [2.0 to 2.7]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is adjusted for multiple comparisons by Hochberg method; Adjusted by level of baseline bone mineral density T-score; Mean Difference (Net) = 2.0, 95% CI 2-sided [1.5 to 2.6] — Denosumab - Placebo

3. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: From Baseline to 12 Months
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 119 | 117
Percent | 0.0 [-0.6 to 0.6] | 2.1 [1.5 to 2.8]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is adjusted for multiple comparisons by Hochberg method; Adjusted by level of baseline bone mineral density T-score; Mean Difference (Net) = 2.2, 95% CI 2-sided [1.3 to 3.0] — Denosumab - Placebo

4. Secondary Outcome: Trochanter Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: From Baseline to 12 Months
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 119 | 117
Percent | 0.8 [0.2 to 1.4] | 3.1 [2.5 to 3.7]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is adjusted for multiple comparisons by Hochberg method; Adjusted by level of baseline bone mineral density T-score; Mean Difference (Net) = 2.3, 95% CI 2-sided [1.4 to 3.2] — Denosumab - Placebo

5. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: From Baseline to 12 Months
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 118 | 116
Percent | -0.3 [-0.8 to 0.2] | 0.6 [0.1 to 1.1]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.0144, ANCOVA — p-value is adjusted for multiple comparisons by Hochberg method; Adjusted by level of baseline bone mineral density T-score; Median Difference (Net) = 0.9, 95% CI 2-sided [0.2 to 1.6] — Denosumab - Placebo

6. Secondary Outcome: Serum Type 1 Collagen C-telopeptide (CTX) Percent Change From Baseline at Day 15
Time Frame: From Baseline to Day 15
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 116 | 115
Percent | -7 [-20 to 16] | -81 [-86 to -75]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, Van Elteren Rank Test — p-value is adjusted for multiple comparisons by Hochberg method; Adjusted by level of baseline bone mineral density T-score

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 10/120 | 11/120
Other Adverse Events (participants affected / at risk) | 27/120 | 23/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | Denosumab 60 mg Q6M (N=120)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Skull malformation (Congenital, familial and genetic disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | Denosumab 60 mg Q6M (N=120)
Constipation (Gastrointestinal disorders) | 7 | 0
Nasopharyngitis (Infections and infestations) | 7 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.